CLINICAL TRIAL: NCT00503880
Title: A Dose Escalation Phase I/II Study of Clofarabine Plus Cytarabine With Growth Factor Priming in Patients Who Are Not Felt to be Candidates for More Aggressive Treatment, With Int-2 and High-Risk MDS
Brief Title: Clofarabine, Cytarabine, and G-CSF in Treating Patients With Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Genzyme discontinued Funding
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0032-07-FB; P30CA036727 (NIH)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Myelodysplastic Syndromes
Keywords: de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Filgrastim; Clofarabine; Cytarabine; Microarray Analysis; Biopsy

ARMS (1):
- Treatment (Experimental): G-CSF 300 μg subcutaneously to begin one day prior to treatment and continued until ANC greater than 1.0 or recovers back to the patients baseline ANC for 3 days in a row subsequent to completion of chemotherapy (SOC) Low-dose Cytarabine 10 mg/m2 subcutaneously daily starting on day 1 for the first 5 consecutive days of the treatment course 2-4 hours following the end of the clofarabine infusion. (SOC) Clofarabine starting at dose level 0. Dose-10 mg/m2 IV over 1 hour daily starting on day 1 for the first 5 consecutive days of the treatment course The G-CSF and cytarabine doses are fixed. The dose of clofarabine is initially fixed. For the subsequent cohort, the dose of clofarabine will be advanced to the next dose level.
  Interventions: Biological: filgrastim; Drug: clofarabine; Drug: cytarabine; Genetic: microarray analysis; Procedure: biopsy

INTERVENTIONS:
Biological: filgrastim — subcutaneously one day prior to treatment
  Other Names: Neupogen
Drug: clofarabine — single IV dose over 1 hour daily for 5 days
  Other Names: Clolar
Drug: cytarabine — subcutaneously daily for 5 days 2-4 hours following the end of the Clofarabine infusion
  Other Names: cytosine arabinoside
Genetic: microarray analysis — Both standard cytogenetic testing and FISH (fluorescent in situ hybridization) are adequate to assess responses.
Procedure: biopsy — bone marrow biopsy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as G-CSF, may increase the number of immune cells found in bone marrow or in peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving clofarabine and cytarabine together with G-CSF may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of clofarabine and to see how well it works when given together with cytarabine and G-CSF in treating patients with myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose (MTD) of clofarabine when administered with low-dose cytarabine and filgrastim (G-CSF) in patients with intermediate-2 or high-risk myelodysplastic syndromes (MDS).
* To evaluate efficacy as measured by hematologic response rates in patients who are treated with this novel combination of drugs and who are not candidates for more intensive treatment for intermediate-2 and high-risk MDS.

Secondary

* To assess effects on quality of life of this patient population.
* To assess the time to acute myeloid leukemia transformation or death.
* To assess cytogenetic response rates.
* To assess changes in flow cytometric patterns.

OUTLINE: This is a phase I, nonrandomized, dose-escalation study of clofarabine followed by a phase II study.

* Phase I: Patients receive clofarabine IV over 1 hour and low-dose cytarabine subcutaneously (SC) on days 1-5. Patients also receive filgrastim (G-CSF) SC beginning 1 day prior to the start of chemotherapy and continuing through completion of chemotherapy until blood counts recover. Treatment repeats every 6 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of clofarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive clofarabine at the MTD, cytarabine, and G-CSF as in phase I.

Quality of life is assessed at baseline, prior to course 4, and after completion of study therapy.

Patients undergo bone marrow biopsy at baseline and prior to courses 3, 6, and 8 for evaluation of treatment response. Bone marrow samples are analyzed for myeloblast phenotypic expression profiles, which include the following parameters: percentage of CD34-positive myeloblasts; antigen expression density of CD13, CD34, CD45, and CD117; and aberrant myeloblast expression of CD4, CD11c, CD15, and CD56.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathologic diagnosis of myelodysplastic syndromes
* International Prognostic Scoring System score of intermediate-2 or high-riskFailed or progressed after 1 prior FDA-approved treatment for MDS OR refused the FDA-approved treatment
* Not a candidate for intensive or standard chemotherapy or stem cell transplantation, as determined by the treating physician
* ECOG performance status 0-2
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 3 times ULN
* Creatinine < 2.0 mg/dL
* Fertile patients must use effective contraception

Exclusion Criteria:

* Not pregnant or nursing
* No comorbidity or condition that, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol or that would decrease life expectancy to < 3 months
* No active, serious infection not controlled by oral or IV antibiotics

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-05-07 (Actual); Primary Completion 2009-10-13 (Actual); Study Completion 2009-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori J Maness, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Cohort #1: Clofarabine Dose Level 0: 10mg/m2
- Phase I: Cohort #2: Clofarabine Dose Level +1: 15 mg/m2
- Phase 1: Dose Cohort #3: Clofarabine Level +2: 20mg/m2
- Phase I: Cohort #4: Clofarabine Level +3: 30 mg/m2
- Phase II: Clinical Response: The presence of hematologic response is the outcome of interest in the Phase II component of the study. Clinical Response will include complete response and partial response.
Period: Overall Study
Arm/Group | Phase I: Cohort #1 | Phase I: Cohort #2 | Phase 1: Dose Cohort #3 | Phase I: Cohort #4 | Phase II: Clinical Response
Started | 2 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 69 [68 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Clofarabine (Phase I)
Description: Maximum Tolerated Dose (MTD) is defined to be the dose cohort below which 2 out of 6 patients experience dose limiting toxicities or the highest dose cohort, if 2 limiting toxicities are not observed at any dose cohort. These will be presented as actual rates. Dose limiting toxicity (DLT) will be defined according to oncology standards based on NCI CTC version 2 grading criteria (DLT = > grade 3 non-hematological toxicity or any > 4 hematological toxicity that persists for more than 4 weeks and in the opinion of the investigator is felt not to be due to disease).
Time Frame: 7 months
Population: Not done - Genzyme discontinued Funding
Groups:
- Treatment: G-CSF 300 μg subcutaneously to begin one day prior to treatment and continued until ANC greater than 1.0 or recovers back to the patients baseline ANC for 3 days in a row subsequent to completion of chemotherapy (SOC) Low-dose Cytarabine 10 mg/m2 subcutaneously daily starting on day 1 for the first 5 consecutive days of the treatment course 2-4 hours following the end of the clofarabine infusion. (SOC) Clofarabine starting at dose level 0(Table 1) dose-10 mg/m2 IV over 1 hour daily starting on day 1 for the first 5 consecutive days of the treatment course.
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Primary Outcome: Presence of Hematologic Response (Phase II)
Description: These are measured in patients with pretreatment abnormalities defined as:
  Hemoglobin < 11 g/dL or transfusion dependence [erythroid- E] Platelets less than 100 x 109/L or platelet-transfusion dependence [platelet- P] Absolute neutrophil count (ANC) less than 1.0 x 109/L [neutrophil- N] Pretreatment baseline measures of cytopenias are averages of at least 2 measurements (not influenced by transfusions)- at least 1 week apart.
Time Frame: Following phase I, responses must last at least 8 weeks.
Population: The study only enrolled 2 patients of the planned 30. The two patients enrolled did not complete the research as planned and were not evaluable. The study was closed due to lack of funding support. Data were not collected.
Groups:
- Treatment: G-CSF 300 μg subcutaneously to begin one day prior to treatment and continued until ANC greater than 1.0 or recovers back to the patients baseline ANC for 3 days in a row subsequent to completion of chemotherapy (SOC) Low-dose Cytarabine 10 mg/m2 subcutaneously daily starting on day 1 for the first 5 consecutive days of the treatment course 2-4 hours following the end of the clofarabine infusion. (SOC) Clofarabine starting at dose level 0: dose-10 mg/m2 IV over 1 hour daily starting on day 1 for the first 5 consecutive days of the treatment course.
Arm/Group | Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Assess Quality of Life
Description: To assess effects on quality of life of this patient population (questionnaire).
Time Frame: 7 months
Population: Not done - Genzyme discontinued Funding
Arm/Group | Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Acute Myelooid Leukemia Transformation or Death.
Description: To assess the time to acute myeloid leukemia transformation or death.
Time Frame: 7months
Population: Not done - Genzyme discontinued Funding
Arm/Group | Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Cytogenetic Response Rates
Description: To assess cytogenetic response rates.
Time Frame: 7 months
Population: Not done - Genzyme discontinued Funding
Arm/Group | Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Changes in Flow of Cytometric Patterns.
Description: To assess changes in flow cytometric patterns.
Time Frame: 7 months
Population: Not done - Genzyme discontinued Funding
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=2)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=2)
ANC (Blood and lymphatic system disorders) | 1 (2)
Bacteremia (Blood and lymphatic system disorders) | 1 (1)
Low Hemoglobin (Blood and lymphatic system disorders) | 1 (2)
Low Platelets (Blood and lymphatic system disorders) | 1 (1)
Low WBC (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 2 (4)
Fatigue (General disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Hemorrhage, ocular
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — petechiae
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (2) — pruritis
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — mental status change
General disorders and administration site conditions (General disorders) | 1 (3) — rash
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — right facial droop
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Right knee pain and swelling
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
White blood cell decreased (Investigations) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) — Angina
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Heartburn

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No